CLINICAL TRIAL: NCT01971723
Title: The Impact of T+ Supplementation on Anabolic Hormone Profile and Performance in Power Athletes
Brief Title: Multi-ingredient Supplement for Strength and Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC#: 2013.10364
Record Dates: First submitted 2013-08-27; First posted 2013-10-29 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Supplement
Keywords: Testosterone; Estrogen; Insulin; Blood Lipid; Glucose; Creatine Kinase; Strength; Power Athlete
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T+ Supplement (Active Comparator): This arm requires the participants to take a prescribed dose of the T+ supplement for 4 weeks while completing an exercise regiment.
  Interventions: Other: T+ Supplement
- Placebo (Placebo Comparator): This arm requires the participants to take a prescribed dose of a calorie matched placebo for 4 weeks while completing an exercise regiment.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: T+ Supplement — Randomized, placebo-controlled, double blind protocol with two treatment groups (matched by lean body mass). Group 1 will receive the recommended serving of one scoop (11g) of T+ supplement. This serving will be taken 45 minutes before the beginning of working out on an empty stomach (>1 hour after meal). On non-training days, the participants will also take a serving at the same time as on training days. This will continue for four weeks (28 days).
  Arms: T+ Supplement
Other: Placebo — The placebo group will consume a calorie-match placebo in the same manner as the supplement group (one serving 45 minutes prior to work outs on an empty stomach). The placebo group will also follow the same supplementation patterns and workout as their counterparts in the supplement group.
  Arms: Placebo

SUMMARY:
It has been suggested that high amounts of total serum testosterone levels correlate with higher lean body mass, lowered fat mass, greater muscle strength, and faster recovery. These suggestions drive athletes and body builders to find ways to raise their testosterone levels. Many athletes and bodybuilders look to alternative methods to anabolic steroids in order increase their testosterone levels without legal repercussions or physiological side effects. Herbs and other plant extracts have been introduced as a possible source to naturally boost testosterone levels. Research supporting the use of herbs and plant extracts has been shown to be equivocal. However, evidence in studies with hypogonadal men suggests that longjack root may naturally boost testosterone levels.

Onnit Labs, LLC has packaged this supplement (T+) which claims it can naturally boost testosterone and lower estrogen levels and subsequently improve performance. This product is a powder (11g) that is mixed with 16 oz of water and consumed 20 minutes prior to anaerobic workouts, such as high intensity weight training.

T+ is a multi-ingredient supplement that consists of vitamins B5 and B6, magnesium aspartic acid, mucuna pruriens, longjack root, nettle root, red clover luteolin, resveratrol, beta- alanine, branch chain amino acids, L- glutamine, Bioperine, and Fibersol 2.

The active ingredients purported to boost plasma testosterone levels are mucuna pruriens, longjack root, and magnesium aspartic acid. The active ingredients claimed to lower plasma estrogen concentrations are red clover, luteolin, resveratrol and nettle root. All other ingredients (Branch Chain Amino Acids and Beta-Alanine) have been documented to improve exercise performance.

It is hypothesized that there will not be any physiological changes after supplementation of T+. It is also hypothesized that performance will not be affected by the supplementation of T+.

DETAILED DESCRIPTION:
The purpose of this study is to examine the physiological and performance effects of T+ on power athletes.

ELIGIBILITY:
Inclusion Criteria:

* Must be familiar with the three main powerlifting movements (squat, bench and deadlift)
* Must have one month training with a designated strength coach to understand the expectations of the strength coach and movement patterns for performance
* Have no pre-existing musculoskeletal disorders
* Participate in the three-week supplement wash out prior to beginning the experiment (except for basic protein supplements and multivitamins)

Exclusion Criteria:

* Female

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ormsbee, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Kreipke VC, Allman BR, Kinsey AW, Moffatt RJ, Hickner RC, Ormsbee MJ. Impact of Four Weeks of a Multi-Ingredient Performance Supplement on Muscular Strength, Body Composition, and Anabolic Hormones in Resistance-Trained Young Men. J Strength Cond Res. 2015 Dec;29(12):3453-65. doi: 10.1519/JSC.0000000000000995. PMID 26595135

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T+ Supplement | Placebo
Started | 16 | 16
Completed | 14 | 13
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T+ Supplement | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 13 | 27
Height (cm) [Mean (Standard Deviation); unit: cm] | 179.13 (5.57) | 177.64 (4.78) | 178.39 (4.51)
Body Mass (kg) [Mean (Standard Deviation); unit: kg] | 75.89 (10.43) | 79.24 (9.71) | 77.43 (9.85)
BMI(kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 24.73 (2.45) | 25.43 (3.15) | 25.06 (2.90)
Total Strength (kg) [Mean (Standard Deviation); unit: kg] — Total strength was calculated by the summation of all one-repetition maxes (squat + bench + deadlift
  kg | 379 (58.61) | 375.87 (70.07) | 375.87 (61.97)

OUTCOME MEASURES:

1. Primary Outcome: Strength Performance Outcomes
Description: Measurement of one repetition maximums strength for all competition lifts included in a standard, ungeared, powerlifting competition (squat, bench, and deadlift). This testing will take place before the supplementation of either T+ or placebo and at the end of the four-week training period.
  Each measure was only compared within it's own category against the baseline measurement and against that of the other group at the same time point.
Time Frame: Baseline measures and 4 weeks from start of study
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
Kg
  Baseline Squat | 119.48 (24.84) | 120.45 (29.82)
  Post Training Squat | 132.47 (26.72) | 129.37 (28.98)
  Baseline Bench | 102.27 (15.75) | 96.33 (22.01)
  Post Training Bench | 108.44 (16.30) | 100.87 (21.69)
  Baseline Deadlift | 157.79 (23.05) | 169.93 (30.07)
  Post Training Deadlift | 171.59 (22.42) | 169.93 (30.07)
  Baseline Total | 379 (58.61) | 375.87 (70.07)
  Post Training Total | 412.5 (60.17) | 400.17 (75.03)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; This statistical analysis is for the squat one repetition maximum outcomes, only; Test type: Superiority or Other; p = .38, ANOVA; Groups were compared against each other at the two different time points and against themselves at the same time points
Statistical Analysis 2: Comparison: T+ Supplement vs Placebo; This statistical analysis is for the bench press one repetition maximum outcomes, only; Test type: Superiority or Other; p = 0.0001, ANOVA
Statistical Analysis 3: Comparison: T+ Supplement vs Placebo; This statistical analysis is for the deadlift one repetition maximum measures, only; Test type: Superiority or Other; p = .3, ANOVA
Statistical Analysis 4: Comparison: T+ Supplement vs Placebo; This statistical analysis compares the outcomes of the total weight lifted; Test type: Superiority or Other; p = 0.0001, ANOVA

2. Primary Outcome: Insulin Outcomes
Description: Measurements of insulin will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: ulU/ml
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
ulU/ml
  Baseline Levels | 5.70 (3.42) | 5.83 (2.73)
  Mid Training Levels | 5.68 (4.51) | 5.34 (2.39)
  Post Training Levels | 5.52 (2.3) | 6.51 (2.67)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

3. Primary Outcome: Blood Lipid Outcomes
Description: Measurements for blood lipid panels will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
mg/dl
  Cholesterol Baseline | 158 (28) | 162 (31)
  Cholesterol Mid Training | 161 (26) | 160 (29)
  Cholesterol Post Training | 162 (27) | 161 (26)
  Glucose Baseline | 93 (11) | 98 (12)
  Glucose Mid Training | 96 (6) | 94 (14)
  Glucose Post Training | 97 (9) | 96 (11)
  HDL Basline | 47 (8) | 50 (8)
  HDL Mid Training | 47 (8) | 50 (9)
  HDL Post Training | 47 (7) | 53 (9)
  LDL Basline | 91 (20) | 91 (27)
  LDL Mid Training | 90 (22) | 86 (21)
  LDL Post Training | 89 (20) | 86 (19)
  Triglycerides Basline | 102 (51) | 88 (38)
  Triglycerides Mid Training | 111 (34) | 94 (37)
  Triglycerides Post Training | 122 (51) | 99 (45)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; This statistical measurement is for cholesterol measure outcomes, only; Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 2: Comparison: T+ Supplement vs Placebo; This statistical analysis is for glucose measure outcomes, only; Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 3: Comparison: T+ Supplement vs Placebo; This statistical analysis is for HDL measure outcomes, only; Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 4: Comparison: T+ Supplement vs Placebo; This statistical analysis is for LDL measure outcomes, only; Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 5: Comparison: T+ Supplement vs Placebo; This statistical analysis for the triglyceride measure outcomes, only; Test type: Superiority or Other; p > .05, ANOVA

4. Primary Outcome: Total Testosterone Outcomes
Description: Measurements for testosterone will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
ng/dL
  Pre Training Levels | 564 (146) | 473 (129)
  Mid Training Levels | 525 (116) | 415 (90)
  Post Training Levels | 548 (148) | 475 (129)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

5. Primary Outcome: Estrogen Outcomes
Description: Measurements for estrogen will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
pg/ml
  Pre Training Levels | 32.7 (16.6) | 31.9 (13.4)
  Mid Training Levels | 33.2 (12.7) | 35.1 (16.1)
  Post Training Levels | 37.4 (12.2) | 35.5 (11.3)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

6. Primary Outcome: Insulin-like Growth Factor-I Outcomes
Description: Measurements for insulin-like growth factor-I will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
ng/dL
  Pre Training Levels | 166 (69) | 213 (74)
  Mid Training Levels | 157 (59) | 207 (67)
  Post Training Levels | 163 (54) | 237 (105)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

7. Primary Outcome: Bio-availableTestosterone Outcomes
Description: Measurements for total testosterone will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
ng/dL
  Pre Training Levels | 321 (105) | 282 (93)
  Mid Training Levels | 286 (91) | 234 (53)
  Post Training Levels | 313 (117) | 273 (90)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

8. Primary Outcome: Free Testosterone Outcomes
Description: Measurements for free testosterone will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
ng/dL
  Pre Training Levels | 13.7 (4.5) | 12.0 (3.9)
  Mid Training Levels | 12.2 (3.9) | 10.0 (2.3)
  Post Training Levels | 13.4 (5.0) | 11.6 (3.8)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

9. Primary Outcome: Dihydrotestosterone Outcomes
Description: Measurements for dihydrotestosterone (DHT) will occur on three occasions: prior to the start of supplementation and training, at the end of two weeks, and finally at the end of training.
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
ng/dL
  Pre Training Levels | 901 (267) | 919 (424)
  Mid Training Levels | 690 (226) | 939 (405)
  Post Training Levels | 926 (427) | 952 (341)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, Chi-squared

10. Secondary Outcome: Volume Performance Outcomes
Description: During the four weeks, the volume ((weight x reps)set 1+(weight x reps)set 2+ (weight x reps)set 3….. ) will be calculated and measured for each exercise in each lifting session.
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: Repetitions
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
Repetitions
  Deadlift | 32.2 (7.7) | 29.9 (8.1)
  Auxiliary Squat | 33.1 (2.5) | 31.5 (4.9)
  Squat | 28 (5.7) | 26 (5.8)
  Bench | 27.4 (6.7) | 26.2 (5.5)
  Total Squat | 30.6 (5.1) | 28.8 (6.0)
  Total Weight Lifted | 30.2 (6.5) | 28.4 (6.6)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; This statistical analysis is for deadlift volume measure outcomes, only; Test type: Superiority or Other; p > .05, t-test, 2 sided
Statistical Analysis 2: Comparison: T+ Supplement vs Placebo; This statistical analysis is for auxiliary squat volume measure outcomes, only; Test type: Superiority or Other; p > .05, t-test, 2 sided
Statistical Analysis 3: Comparison: T+ Supplement vs Placebo; This statistical analysis is for squat volume measure outcomes, only; Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 4: Comparison: T+ Supplement vs Placebo; This statistical analysis is for bench volume measure outcomes, only; Test type: Superiority or Other; p > .05, t-test, 2 sided
Statistical Analysis 5: Comparison: T+ Supplement vs Placebo; This statistical analysis is for total squat volume measures, only; Test type: Superiority or Other; p > .05, t-test, 2 sided
Statistical Analysis 6: Comparison: T+ Supplement vs Placebo; This statistical analysis is for total weight lifted volume measure outcomes, only; Test type: Superiority or Other; p > .05, t-test, 2 sided

11. Primary Outcome: Cortisol Outcomes
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
ug/dl
  Pre Training Levels | 17.0 (4.1) | 20.1 (4.0)
  Mid Training Levels | 17.7 (4.4) | 19.9 (3.9)
  Post Training Levels | 19.3 (3.1) | 19.2 (3.0)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

12. Primary Outcome: Sex-hormone Binding Globulin Outcomes
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
nmol/l
  Pre Training Levels | 28.2 (12.3) | 23.5 (10.4)
  Mid Training Levels | 32.0 (14.4) | 25.5 (11.0)
  Post Training Levels | 30.3 (13.8) | 26 (11.6)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p > .05, ANOVA

13. Primary Outcome: Creatine-Kinase Outcomes
Time Frame: Baseline, 2-week mark, 4-week mark
Measure: Mean (Standard Deviation); unit: mkat/L
Arm/Group | T+ Supplement | Placebo
Number analyzed (Participants) | 14 | 13
mkat/L
  Pre Training Levels | 2.0 (1.0) | 2.2 (2.4)
  Mid Training Levels | 2.5 (1.7) | 1.7 (0.9)
  Post Training Levels | 1.8 (1.2) | 1.8 (1.7)
Statistical Analysis 1: Comparison: T+ Supplement vs Placebo; Test type: Superiority or Other; p = .05, ANOVA

ADVERSE EVENTS:
Time Frame: Reports were only collected during the 4 weeks of training.
Arm/Group | T+ Supplement | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 5/14 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T+ Supplement (N=14) | Placebo (N=13)
Increased Libido (Reproductive system and breast disorders) | 2 (2) | 0 — Subjects reported increased libidos
paresthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Tingling of the skin
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Subjects reported more acne than usual

LIMITATIONS AND CAVEATS:
Unable to standardize individual ingredients in T+ supplement. Volume of lifts not tested was not analyzed for statistical significance. Neuromuscular adaptations were not tested. Length of study may have affected body composition measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No